CLINICAL TRIAL: NCT00872066
Title: A Prospective, Randomised, Uncontrolled, Single-Centre, Post-Market Surveillance Study To Evaluate The Performance Of SmartSet® HV and SmartSet® GHV Bone Cements In Primary Cemented Total Hip Arthroplasty(THA)
Brief Title: A Study to Assess the Long-term Performance of SmartSet® HV and SmartSet® GHV Bone Cements in Primary Total Hip Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT02/11
Record Dates: First submitted 2009-03-19; First posted 2009-03-31 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Traumatic Femoral Fractures; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Bone Cement
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1) SmartSet® HV Bone Cement (Active Comparator): A high viscosity bone cement for use in total hip replacement (without gentamicin)
  Interventions: Device: SmartSet® HV bone cement
- 2) SmartSet® GHV Bone Cement (Active Comparator): A high viscosity bone cement for use in total hip replacement (with gentamicin)
  Interventions: Device: SmartSet® GHV bone cement

INTERVENTIONS:
Device: SmartSet® HV bone cement — A high viscosity bone cement for use in total hip replacement (without gentamicin)
  Arms: 1) SmartSet® HV Bone Cement
Device: SmartSet® GHV bone cement — A high viscosity bone cement for use in total hip replacement (with gentamicin)
  Arms: 2) SmartSet® GHV Bone Cement

SUMMARY:
The purpose of this study is to monitor the performance of artificial hip joints implanted with two different bone cements, SmartSet® HV and SmartSet® GHV, in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be randomly allocated to SmartSet® HV or SmartSet® GHV and will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged between 18 and 75 years (inclusive).

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects requiring primary total hip arthroplasty and are considered suitable for a cemented femoral component.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.

ii) Women who are pregnant.

iii) Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.

iv) Subjects who have participated in a clinical study with an investigational product in the last 6 month(s).

v) Subjects who are currently involved in any injury litigation claims.

vi) Subjects with contraindications normally applicable to the use of conventional bone cement, in accordance with the manufacturer's Instructions For Use.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2006-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Kaplan-Meier survivorship | Annually

SECONDARY OUTCOMES:
Harris Hip Score | Annually
Oxford Hip Score | Annually
Radiological Analysis | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Libor Nečas, M.D., Principal Investigator — Orthopaedic-truamatology Clinic, University Hospital Martin, Slovakia
Locations (1):
- Orthopaedic-traumatology Clinic University Hospital Martin, Martin, Slovakia